CLINICAL TRIAL: NCT00757107
Title: Clinical Evaluation of Taperloc Total Hip System With Two Different Stem Lengths
Brief Title: Taperloc Versus Taplerloc Microplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingemar Ivarsson (Other)
Collaborators: Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Ingemar Ivarsson, Associate Professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMET.CR.ROWEU1
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Short femoral stem; Stress shielding; Stem migration; Implant Survival; DEXA; Radiostereometric analysis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taperloc Microplasty (Experimental): Patients with primary osteoarthritis with Taperloc microplasty non inferiority
  Interventions: Device: Taperloc Microplasty
- Taperloc Standard (Active Comparator): Patients with primary osteoarthritis Taperloc standard
  Interventions: Device: Taperloc standard

INTERVENTIONS:
Device: Taperloc Microplasty — primary total hip arthroplasty
  Arms: Taperloc Microplasty
Device: Taperloc standard — primary total hip arthroplasty
  Arms: Taperloc Standard

SUMMARY:
This evaluation is conducted to evaluate the safety and performance of two different stem lengths of the Taperloc Total Hip System. Per implant bone loss and migration of the stem are compared between the two groups with Dual-energy X-ray absorptiometry (DEXA) and radiostereomektric analysis

DETAILED DESCRIPTION:
Consecutive patients between 50 - 70 years diagnosed with primary osteoarthritis of the hip and eligible for total hip arthroplasty will be asked to participate in the study.

Periprosthetic bone loss, migration of the components and clinical scores will be recorded prospectively at 3,6,12 and 24 months.

ELIGIBILITY:
Inclusion criteria:

* Patients with primary osteoarthritis of the hip scheduled for THA.
* Suitable anatomy for both stems
* Willingness and ability to follow study-protocol

Exclusion Criteria

* Malignancy or metastatic bone disease.
* Any other disease severely affecting bone and mineral metabolism
* Ongoing or previous treatment (within 5 years prior to inclusion) with steroids
* Ongoing or previous treatment (within 5 years prior to inclusion) with antiresorptives.
* Ongoing or previous treatment (within 5 years prior to inclusion) with immunosuppressive drugs.
* Ongoing or previous treatment (within 5 years prior to inclusion) with anticonvulsive therapy.
* Ongoing or previous treatment (within 5 years prior to inclusion) with hormonal therapy.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Bone remodelling, i e change in bone mineral density around the stem, as measured with dual energy x-ray absorptiometry (DEXA) [ Time Frame: | bone mineral density (BMD) measured postoperatively at 2 years

SECONDARY OUTCOMES:
Migration of stem components in six degrees of freedom and maximum total point motion measured with radiostereometric analysis | 2 years

OTHER OUTCOMES:
Clinical outcome measures with Harris Hip Score comparing patients receiving different stems. | 3, 6, 12 and 24 months
Clinical outcome measures with Womac Score comparing patients receiving different stems. | 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar IVARSSON, PhD, Principal Investigator — University hospital of Linkoping
Locations (1):
- University hospital of Linkoping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes